CLINICAL TRIAL: NCT03407326
Title: Comparison of an Alternative Therapeutic Food for the International Food Aid Market to a Standard Ready-to-use Therapeutic Food (RUTF) for the Treatment of Severe Acute Malnutrition in Children of the Western Rural Region and Pujehun District of Sierra Leone
Brief Title: Comparison of an Alternative Therapeutic Food for the International Food Aid Market to a Standard Ready-to-use Therapeutic Food (RUTF) for the Treatment of Severe Acute Malnutrition in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: The Children's Investment Fund Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 201710147
Record Dates: First submitted 2018-01-16; First posted 2018-01-23 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Malnutrition
Keywords: severe acute malnutrition, SAM
MeSH Terms: conditions — Malnutrition; Severe Acute Malnutrition

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alternative (Experimental): Participants will receive approximately 190 kcal/kg/day of alternative RUTF till recovery or up to 12 weeks of treatment.
  Interventions: Dietary Supplement: Alternative RUTF
- Standard (Active Comparator): Participants will receive approximately 190 kcal/kg/day of standard RUTF till recovery or up to 12 weeks of treatment.
  Interventions: Dietary Supplement: Standard RUTF

INTERVENTIONS:
Dietary Supplement: Alternative RUTF — The alternative RUTF contains oat, peanuts, sugar, milk powder, vegetable oil as well as premix containing concentrated minerals and vitamins and emulsifier.
  Arms: Alternative
Dietary Supplement: Standard RUTF — Standard RUTF contains peanut paste, sugar, non-fat dried milk (NFDM), vegetable oil, a premix containing concentrated minerals and vitamins, and emulsifier.
  Arms: Standard

SUMMARY:
In this clinical non-inferiority trial, two foods will be compared for the treatment of SAM, testing the hypothesis that the difference in recovery rates and growth between the two test groups will be no greater than 5 percent.

DETAILED DESCRIPTION:
This will be a randomised, triple-blinded, controlled clinical non-inferiority trial assessing the treatment of SAM with one of two therapeutic foods until the child is recovered or for a period of up to 12 weeks.

Subjects will be recruited from rural health clinics in the Western Rural Region and Pujehun District of Sierra Leone, due to the limited accessibility of treatment programs in this area; investigators believe a clinical trial in this district will be beneficial.

Sierra Leonean children aged 6-59 months with uncomplicated SAM (with WHZ < -3, MUAC of <11.5 cm, or bipedal edema) will be recruited at health clinics in the Western Rural Region and Pujehun District. A total of 1,300 children will be enrolled for a total sample size of 1,262 (631 per treatment) from 30 PHU centers, to detect a 5% difference in recovery rates between any two foods, with 95% sensitivity and 80% power, assuming that the standard recovery rate is 85% and a binary non-inferiority test.

After screening and enrolment, each child's participation will last up to 12 weeks. If a child recovers before the end of the 12-week period, a child's WHZ reaches and stays above -2 for two consecutive visits without edema, the child will graduate from the study. No study food products will be given to children after 12 weeks of participation; those who have not recovered will be taken for inpatient treatment. Children will enter the study on a rolling enrolment basis and will continue to be enrolled until 1,300 children complete the study.

Random allocation of food intervention will be conducted by nurses who will have the caregiver draw opaque envelopes containing one of 4 colours. Caretakers chose a sealed envelope that contains 1 of 4 colours: 2 of these colours correspond to the control food and 2 to the experimental food. The colour will be recorded separately from the child's clinical measurements and researchers involved in the randomization process do not know which colour corresponds to which food corresponding to one of the therapeutic foods. The code will be accessible only to the food distribution personnel, who do not assess participant outcomes or eligibility. Investigators performing clinical assessments and caretakers will be blinded to the child's assigned food group.

A sub-set of participants in the main study will undergo eye-tracking testing to evaluate neurocognitive function and recovery in children with severe acute malnutrition after receiving therapeutic food.

ELIGIBILITY:
Inclusion Criteria: Children aged 6-59 months with one or combination of the following

* WHZ < -3
* MUAC <11.5cm
* bipedal edema

Exclusion Criteria:

* children currently involved in another research trial or feeding program
* developmentally delayed
* chronic debilitating illness (such as cerebral palsy)
* history of peanut or milk allergy

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1568 (Actual)
Dates: Start 2018-10-16 (Actual); Primary Completion 2019-09-02 (Actual); Study Completion 2019-09-02 (Actual)

PRIMARY OUTCOMES:
Mid-upper-arm circumference | 2 to 12 weeks
  MUAC ≥ 12.5
Weight-for-height z score | 2 to 12 weeks
  WHZ≥-2

SECONDARY OUTCOMES:
Adverse symptoms | 2 to 12 weeks
  stomach pain, vomiting, diarrhoea, rash or fever

CONTACTS AND LOCATIONS:
Locations (1):
- Project Peanut Butter, Freetown, Sierra Leone

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hendrixson DT, Godbout C, Los A, Callaghan-Gillespie M, Mui M, Wegner D, Bryant T, Koroma A, Manary MJ. Treatment of severe acute malnutrition with oat or standard ready-to-use therapeutic food: a triple-blind, randomised controlled clinical trial. Gut. 2020 Dec;69(12):2143-2149. doi: 10.1136/gutjnl-2020-320769. Epub 2020 Mar 16. PMID 32179568